CLINICAL TRIAL: NCT03373604
Title: Imaging Tau in Alzheimer's Disease and Normal Aging With 18F-MK-6240
Brief Title: Imaging Tau in Alzheimer's Disease and Normal Aging
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Patrick Lao (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor-Investigator, Patrick Lao, Assistant Professor of Neurological Sciences, Columbia University
Organization: Columbia University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: AAAR4352; K23AG052633-02 (NIH); 2R56AG034189-06A1 (NIH); K24AG045334 (NIH); R01AG055299 (NIH); R01AG050440-02S1 (NIH)
Record Dates: First submitted 2017-12-11; First posted 2017-12-14 (Actual); Results first posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: Alzheimer Disease
Keywords: 18F-MK-6240; Cognitive Impairment; Alzheimer's
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — Spinal Puncture

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cognitive impairment (Experimental): Alzheimer's disease (mild cognitive impairment or mild stage Alzheimer's disease dementia)
  Interventions: Drug: 18F-MK-6240; Procedure: Lumbar Puncture (optional)
- No cognitive impairment (Active Comparator): Healthy controls
  Interventions: Drug: 18F-MK-6240; Procedure: Lumbar Puncture (optional)

INTERVENTIONS:
Drug: 18F-MK-6240 — 18F-MK-6240 is a PET radioligand that binds abnormal tangles made of the protein tau. These tau tangles develop in the brain in people with Alzheimer's disease.
  Other Names: [18F]-MK6240
Procedure: Lumbar Puncture (optional) — Subjects have the option to have lumbar puncture performed for the measurement of Alzheimer's disease biomarkers in cerebrospinal fluid.

SUMMARY:
This study is being done to learn about tau tangles in Alzheimer's disease. A type of positron emission tomography (PET) scan is used to measure the abnormal accumulation of protein called tau in the brain. These are thought to be involved in Alzheimer's disease. The investigators will also perform brain MRI and to tests to measure the participant's memory and thinking.

DETAILED DESCRIPTION:
This study is being done to determine the relationship between tau tangles and cognitive impairment in elderly subjects with and without Alzheimer's disease (AD). Subjects will undergo screen that includes neuropsychological testing and brain MRI. This study uses a special type of scan called a PET scan to take pictures of the brain. During the PET scan, a special radioactive dye called 18F-MK-6240 is injected into the body. 18F-MK-6240 sticks to abnormal tangles made of the protein tau. Subjects will have the option to have lumbar puncture performed to measure CSF concentrations of biomarkers.

ELIGIBILITY:
Inclusion Criteria:

1. Age 50 and older.
2. Meet criteria for either

   1. amnestic mild cognitive impairment (MCI) (single or mixed domain) or mild Alzheimer's disease (AD), or
   2. have no cognitive impairment, based on history, exam, neuropsychological testing, and consensus diagnosis. MCI and mild AD patients must have Clinical Dementia Rating scale score of 0.5 or 1. Unimpaired subjects must have Clinical Dementia Rating scale score of 0.
3. Subjects unable to provide informed consent must have a surrogate decision maker.
4. Written and oral fluency in English or Spanish.
5. Able to participate in all scheduled evaluations and to complete all required tests and procedures.
6. In the opinion of the investigator, the subject must be considered likely to comply with the study protocol and to have a high probability of completing the study.

Exclusion Criteria:

1. Past or present history of certain brain disorders other than MCI or AD.
2. Certain significant medical conditions, which make study procedures of the current study unsafe. Such serious medical conditions include uncontrolled epilepsy and multiple serious injuries.
3. Contraindication to magnetic resonance imaging (MRI) scanning.
4. Conditions precluding entry into the scanners (e.g. morbid obesity, claustrophobia, etc.).
5. History of kidney disease or presence of impaired kidney function based on laboratory tests at screening visit.
6. History of liver disease or presence of impaired liver function based on laboratory tests at screening visit.
7. Participation in the last year in a clinical trial for a disease modifying drug for AD.
8. Inability to have a catheter in subject's vein for the injection of radioligand.
9. Inability to have blood drawn from subject's veins.

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2017-12-11 (Actual); Primary Completion 2022-05-11 (Actual); Study Completion 2022-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Lao, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

REFERENCES:
- [Derived] Klein J, Yan X, Johnson A, Tomljanovic Z, Zou J, Polly K, Honig LS, Brickman AM, Stern Y, Devanand DP, Lee S, Kreisl WC. Olfactory Impairment Is Related to Tau Pathology and Neuroinflammation in Alzheimer's Disease. J Alzheimers Dis. 2021;80(3):1051-1065. doi: 10.3233/JAD-201149. PMID 33646153

RESULTS

PARTICIPANT FLOW:
Groups:
- No Cognitive Impairment: Healthy participants without cognitive impairment
- Cognitive Impairment: Participants with mild cognitive impairment or mild stage Alzheimer's disease dementia
Period: Overall Study
Arm/Group | No Cognitive Impairment | Cognitive Impairment
Started | 43 | 28
Completed | 43 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Cognitive Impairment | Cognitive Impairment | Total
Number analyzed (Participants) | 43 | 28 | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.6 (8.6) | 69.5 (10.2) | 70.1 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 7 | 28
  Male | 22 | 21 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 40 | 26 | 66
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 16 | 2 | 18
  White | 27 | 26 | 53
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 43 | 28 | 71

OUTCOME MEASURES:

1. Primary Outcome: 18F-MK-6240 Binding
Description: Standardized uptake value ratio (SUVr)
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: SUVr
Arm/Group | No Cognitive Impairment | Cognitive Impairment
Number analyzed (Participants) | 43 | 28
SUVr | 1.41 (0.43) | 2.30 (0.92)

2. Secondary Outcome: Correlation Between Tau, Neurodegeneration and Inflammation Using PET and CSF Biomarkers.
Description: Correlation of 18F-MK-6240 binding and CSF markers of neurodegeneration and inflammation.
Time Frame: One year follow-up
Measure: Number; unit: correlation coefficient (r)
Arm/Group | No Cognitive Impairment | Cognitive Impairment
Number analyzed (Participants) | 43 | 28
correlation coefficient (r)
  Correlation between Tau and Neurodegeneration | -0.347 | 0.013
  Correlation between Tau and Inflammation | -0.295 | 0.181

ADVERSE EVENTS:
Time Frame: During the scanning procedure (1 day), and at 1 year follow-up
Arm/Group | No Cognitive Impairment | Cognitive Impairment
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/28
Other Adverse Events (participants affected / at risk) | 4/43 | 4/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | No Cognitive Impairment (N=43) | Cognitive Impairment (N=28)
Sore arm from IV placement (Injury, poisoning and procedural complications) | 0 | 1
Elevated blood pressure (Blood and lymphatic system disorders) | 1 | 1
hypoglycemia (Blood and lymphatic system disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
lightheadedness (General disorders) | 1 | 0
musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-21): https://cdn.clinicaltrials.gov/large-docs/04/NCT03373604/Prot_SAP_000.pdf